CLINICAL TRIAL: NCT00657501
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study of the Safety and Efficacy of LibiGel® for the Treatment of Hypoactive Sexual Desire Disorder in Surgically Menopausal Women
Brief Title: Safety and Efficacy of LibiGel® for Treatment of Hypoactive Sexual Desire Disorder in Surgically Menopausal Women
Acronym: BLOOM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioSante Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TESTW008
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: testosterone; hypoactive sexual desire disorder; menopause
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Testosterone Propionate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- testosterone gel (Experimental): 1% testosterone transdermal gel
  Interventions: Drug: testosterone gel
- Placebo gel (Placebo Comparator): placebo transdermal gel
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: testosterone gel — once daily transdermal gel, 300 mcg
  Other Names: LibiGel
  Arms: testosterone gel
Drug: placebo gel — once daily transdermal placebo gel
  Arms: Placebo gel

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, multi-center study of the safety and efficacy of LibiGel 300mcg in the treatment of HSDD in surgically menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 30 to 65 years
* Must have undergone hysterectomy and bilateral salpingo-oophorectomy

Exclusion Criteria:

* A history of allergic reactions to androgens (oral or patch), topical alcohol, or any component of the formulation
* Any systemic skin diseases or local skin abnormalities in the area of application
* Diagnosed with another primary female sexual dysfunction (e.g., Sexual Aversion Disorder, Female Sexual Arousal Disorder).
* A medical condition that could affect or interfere with sexual function
* Using a systemic transdermal gel or cream estrogen therapy.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Co-primary endpoints are the change in the 4-week total number of satisfying sexual events from the Baseline period to Weeks 21-24, and the change from Baseline to Weeks 21-24 in the mean ISED desire score. | Time Frame: Baseline and 21-24 weeks.

SECONDARY OUTCOMES:
Change from baseline over time for multiple efficacy measurements | change over timepoints from baseline period

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Snabes, MD, PhD, Study Director — BioSante Pharmaceuticals, Inc.
Locations (69):
- United States (66):
  - BioSante Site #146, Mobile, Alabama
  - BioSante Site #171, Chandler, Arizona
  - BioSante Site #145, Glendale, Arizona
  - BioSante Site #121, Phoenix, Arizona
  - BioSante Site #137, Tucson, Arizona
  - BioSante Site #100, Jonesboro, Arkansas
  - BioSante Site #155, Little Rock, Arkansas
  - BioSante Site #221, Berkely, California
  - BioSante Site #162, Sacramento, California
  - BioSante Site #112, San Diego, California
  - BioSante Site #159, Walnut Creek, California
  - BioSante Site #026, Lakewood, Colorado
  - BioSante Site #166, Farmington, Connecticut
  - BioSante Site #132, New Britain, Connecticut
  - BioSante Site #151, New London, Connecticut
  - BioSante Site #143, Jacksonville, Florida
  - BioSante Site #111, Orlando, Florida
  - BioSante Site #152, Tampa, Florida
  - BioSante Site #115, Atlanta, Georgia
  - BioSante Site #141, Roswell, Georgia
  - BioSante Site #202, Idaho Falls, Idaho
  - BioSante Site #017, Meridian, Idaho
  - BioSante Site #156, Champaign, Illinois
  - BioSante Site #045, Chicago, Illinois
  - BioSante Site #149, Chicago, Illinois
  - BioSante Site #133, Chicago, Illinois
  - BioSante Site #167, Newburgh, Indiana
  - BioSante Site #163, Overland Park, Kansas
  - BioSante Site #214, Lexington, Kentucky
  - BioSante Site #136, Lexington, Kentucky
  - BioSante Site #157, Mandeville, Louisiana
  - BioSante Site #110, Metarie, Louisiana
  - BioSante Site #035, Ann Arbor, Michigan
  - BioSante Site #124, Bingham Farms, Michigan
  - BioSante Site #105, Kalamazoo, Michigan
  - BioSante Site #104, St Louis, Missouri
  - BioSante Site #127, Billings, Montana
  - BioSante Site #114, Las Vegas, Nevada
  - BioSante Site #161, Purchase, New York
  - BioSante Site #107, Raleigh, North Carolina
  - BioSante Site #131, Winston-Salem, North Carolina
  - BioSante Site #130, Beachwood, Ohio
  - BioSante Site #101, Cleveland, Ohio
  - BioSante Site #160, Englewood, Ohio
  - BioSante Site #153, Gallipolis, Ohio
  - Site #170, Kettering, Ohio
  - BioSante Site #116, Mayfield Heights, Ohio
  - BioSante Site #138, West Chester, Ohio
  - BioSante Site #129, Tulsa, Oklahoma
  - BioSante Site #106, Eugene, Oregon
  - BioSante Site #126, Medford, Oregon
  - BioSante Site #203, Portland, Oregon
  - BioSante Site #165, Jenkintown, Pennsylvania
  - BioSante Site #142, Pittsburgh, Pennsylvania
  - BioSante Site #099, Sellersville, Pennsylvania
  - BioSante Site #075, Warwick, Rhode Island
  - BioSante Site #117, Anderson, South Carolina
  - BioSante Site #120, North Jackson, Tennessee
  - BioSante Site #147, Dallas, Texas
  - BioSante Site #122, Houston, Texas
  - BioSante Site #154, Hurst, Texas
  - BioSante Site #084, San Antonio, Texas
  - BioSante Site #144, Pleasant Grove, Utah
  - BioSante Site #102, Salt Lake City, Utah
  - BioSante Site #128, Seattle, Washington
  - BioSante Site #183, Walla Walla, Washington
- Canada (3):
  - BioSante Site #175, Vancouver, British Columbia
  - BioSante Site #123, Ottawa, Ontario
  - BioSante Site #109, Québec, Quebec

REFERENCES:
- See also: Bloomstudy.com — http://www.bloomstudy.com